CLINICAL TRIAL: NCT04256746
Title: A Natural Extract for Reducing the Post Prandial Blood Glucose Response in Healthy Indian Adults: A Dose-response Study of Efficacy and Tolerance
Brief Title: Dose Response Study of a Natural Extract for Reducing Post Prandial Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Lambda Therapeutic Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-NAA-0720
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Blood Glucose

STUDY DESIGN:
Intervention Model Description: Randomized, balanced incomplete block design dose response study of efficacy,
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The coded and un-coded randomization schedule was generated by the bio-statistician of CRO.
  The person involved in the preparation of the test product was not involved in any other activities related to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Boiled Rice (Placebo Comparator): 63 g of raw rice was cooked.
  Interventions: Other: Boiled Rice
- Boiled Rice+0.37 gr extract (Experimental): 63 g of raw rice was cooked and 0.37 gr mulberry fruit powdered extract added and mixed
  Interventions: Other: Boiled Rice+0.37 gr mulberry fruit powdered extract
- Boiled Rice+0.75 gr extract (Experimental): 63 g of raw rice was cooked and 0.75 gr mulberry fruit powdered extract added and mixed
  Interventions: Other: Boiled Rice+0.75 gr mulberry fruit powdered extract
- Boiled Rice+1.12 gr extract (Experimental): 63 g of raw rice was cooked and 1.12 gr mulberry fruit powdered extract added and mixed
  Interventions: Other: Boiled Rice+1.12 gr mulberry fruit powdered extract
- Boiled Rice+1.50 gr extract (Experimental): 63 g of raw rice was cooked and 1.50 gr mulberry fruit powdered extract added and mixed
  Interventions: Other: Boiled Rice+1.50 gr mulberry fruit powdered extract
- Rice porridge (Placebo Comparator): 60 g of rice porridge was rehydrated with 300 ml boiling hot water
  Interventions: Other: Rice Porridge
- Rice porridge+1.50 gr extract (Active Comparator): 60 g of rice porridge was rehydrated with 300 ml boiling hot water and 1.50 gr mulberry fruit powdered extract added and mixed
  Interventions: Other: Rice porridge+1.50 gr mulberry fruit powdered extract

INTERVENTIONS:
Other: Boiled Rice
  Arms: Boiled Rice
Other: Boiled Rice+0.37 gr mulberry fruit powdered extract
  Arms: Boiled Rice+0.37 gr extract
Other: Boiled Rice+0.75 gr mulberry fruit powdered extract
  Arms: Boiled Rice+0.75 gr extract
Other: Boiled Rice+1.12 gr mulberry fruit powdered extract
  Arms: Boiled Rice+1.12 gr extract
Other: Boiled Rice+1.50 gr mulberry fruit powdered extract
  Arms: Boiled Rice+1.50 gr extract
Other: Rice Porridge
  Arms: Rice porridge
Other: Rice porridge+1.50 gr mulberry fruit powdered extract
  Arms: Rice porridge+1.50 gr extract

SUMMARY:
Randomized, balanced incomplete block design dose response study of efficacy, with 4 different dosages of mulberry fruit powdered extract added to cooked rice compared to a reference treatment (cooked rice only).

DETAILED DESCRIPTION:
Dose response study with 4 dosages of mulberry fruit powdered extract (0.37, 0.75, 1.12 and 1.5 g) added to cooked rice, compared to cooked rice only(reference) on post prandial blood glucose response in healthy Indian adults.

In addition, 1.5 g of mulberry fruit powdered extract was added to instant rice porridge and compared to instant rice porridge only as positive control (replication of previous research.

In total there were 7 test products in the study: 5 active treatments and 2 reference treatments.

The study was a cross-over study (4 interventions per subject, 4 out of the 7 test products). The recovery period between treatments was at least seven days.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give consent to participate in the study in writing;
* Healthy male and female subjects between ≥ 20 and ≤ 50.0 years of age;
* BMI of ≥18.0 and ≤ 25.0 kg/m2;
* Apparently healthy: no medical conditions which might effect study measurements as judged by the study physician or measured by questionnaire, and/or assessed by hematology, blood chemistry and urinalysis;
* Willing to comply to study protocol during the study;
* Agreeing to be informed about medically relevant personal test-results by study physician;
* Willing to refrain from drinking of alcohol on and one day before the blood withdrawal;
* Fasting blood glucose value of volunteer is ≥ 3.4 and ≤ 6.1 mmol/litre (i.e. 62-110 mg/dl) at screening;
* Haemoglobin level within clinically acceptable range (for male 12 to 17 gm/dL and for females 11 to 15 gm / dL; both inclusive) as judged by the research physician.

Exclusion Criteria:

* Being an employee of Unilever of Lambda;
* Chronic smokers, tobacco chewers and drinkers;
* Participation in any other biomedical study 3 months before screening visit day of this study and/or participating in any other biomedical study during the screening period;
* High intake of alcohol (>120 mL/week);
* Reported use of medically prescribed/slimming diet;
* Reported participation in night shifts (between 23.00 and 6.00 hrs);
* Use of medication which interferes with study measurements including vitamins, tonics;
* Reported intense exercise ≥10 h/week;
* Reported weight loss/gain ≥ 10% of body weight in the 6 months preceding screening
* Blood donation for 2 months prior to screening;
* Urine analysis that showed any drug abuse;
* Allergy to any food or cosmetics;
* If female, not being pregnant or planning pregnancy during the study period;
* If female, lactating or has been lactating for 6 weeks before pre-study investigation and/or during the study period.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2012-09-24 (Actual); Primary Completion 2012-10-19 (Actual); Study Completion 2012-10-19 (Actual)

PRIMARY OUTCOMES:
Post-prandial blood glucose | Positive incremental Area under the glucose versus time Curve between 0 (before) and 2 hours after test product intake
  Glucose concentration in venous plasma

SECONDARY OUTCOMES:
Post-prandial insulin | Total area under the insulin versus time curves between 0 (before) and 2 hours after study product intake
  Post-prandial serum insulin

OTHER OUTCOMES:
Hydrogen gas in exhaled breath | Analyzed before study product administration at 20 minutes before and at 65, 125, 185, 245, 305, 365 and 425 minutes after the ingestion of the study products
  Each time a volunteer produced a 10 ppm hydrogen (or more) above the basal breath hydrogen level during the 7-hour test period, the value was regarded as a "positive".
Intestinal discomfort | Just before and at 430 minutes after study product administration
  A questionnaire to assess four aspects of intestinal discomfort (bloating, flatulence, nausea and pain) on scale from 0-3 was completed by the subjects

CONTACTS AND LOCATIONS:
Overall Officials: David Mela, Dr., Study Director — Unilever R&D Vlaardingen (retired)
Locations (1):
- Lambda Therapeutics Research Ttd (LTRL), Ahmedabad, Gujarat, India